CLINICAL TRIAL: NCT05647564
Title: PET/CT Characterization of Treatment Resistance of AR-targeted Therapies in mCRPC
Brief Title: PET/CT Characterization of Treatment Resistance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-0910; 2022-0910 (Other: UW Madison); A534260 (Other: UW Madison); SMPH/MEDICINE/HEM-ONC (Other: UW Madison); NCI-2022-09580 (Registry Identifier: NCI); Protocol Version 3/22/2024 (Other: UW Madison)
Record Dates: First submitted 2022-12-06; First posted 2022-12-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: androgen receptor targeted therapy; imaging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrinsic Resistance Cohort (Cohort A) (Other): Participants assigned to Cohort A have advanced prostate cancer and are scheduled to start a second-generation AR-targeted (such as enzalutamide, abiraterone, darolutamide, or apalutamide) or PSMA directed (e.g. Lu177-PSMA) therapies .
  Interventions: Diagnostic Test: F-fluorodeoxyglucose positron emission tomography (FDG PET); Diagnostic Test: prostate-specific membrane antigen positron emission tomography (PSMA PET)
- Acquired Resistance Cohort (Cohort B) (Other): Participants are assigned to Cohort B if they have advanced prostate cancer, are already on a second-generation AR-targeted therapy, and have shown an increase in their PSA (prostate-specific antigen) levels.
  Interventions: Diagnostic Test: F-fluorodeoxyglucose positron emission tomography (FDG PET); Diagnostic Test: prostate-specific membrane antigen positron emission tomography (PSMA PET)

INTERVENTIONS:
Diagnostic Test: F-fluorodeoxyglucose positron emission tomography (FDG PET) — Imaging scan
Diagnostic Test: prostate-specific membrane antigen positron emission tomography (PSMA PET) — Imaging scan

SUMMARY:
This study will use different types of medical imaging to assess how lesions from advanced prostate cancer become resistant to second-generation AR-targeted therapy, and how the different types of imaging compare in that assessment. Participants in this study have advanced prostate cancer and are either scheduled to start a second-generation androgen receptor (AR) targeted therapy (such as enzalutamide, abiraterone, or apalutamide) or are already being treated with one. Participants can expect to be in the study for at least 9 months, and up to 2 years.

DETAILED DESCRIPTION:
There are two groups, or cohorts, in this study. Participants are assigned to Cohort A if they have advanced prostate cancer and are scheduled to start a second-generation AR-targeted therapy (such as enzalutamide, abiraterone, darolutamide, or apalutamide) or PSMA directed radiotherapy (e.g. Lu177-PSMA radio-ligand therapy. Participants are assigned to Cohort B if they have advanced prostate cancer, are already on a second-generation AR-targeted therapy, and have shown an increase in their PSA (prostate-specific antigen) levels.

There are two medical imaging scans that will be done for research purposes in this study. One is called 18F-fluorodeoxyglucose positron emission tomography (FDG PET) and the other is prostate-specific membrane antigen positron emission tomography (PSMA PET). These scans are done simultaneously with computed tomography (CT) scanning. Participants will be scheduled to have 6 scans, 3 FDG PET/CT scans and 3 PSMA PET/CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate.
* At least 1 radiographic metastases as seen on conventional CT imaging or bone scan
* Progressive prostate cancer as evident by at least two separate increase in PSA over nadir, and absolute PSA value at least 2 ng/ml (INTRINSIC RESISTANCE COHORT ONLY)
* Patients must be candidate for a second-generation androgen receptor (AR) inhibitor (e.g. enzalutamide, abiraterone, darolutamide, apalutamide), or Lu177-PSMA radioligand therapy (INTRINSIC RESISTANCE COHORT ONLY)
* Men of age >18 years.
* Patients must be able to comply with all study procedures, including having both the ability and willingness to lie flat for ≥ 30 minutes during imaging
* Patients must be informed of the exploratory nature of the study and its potential risks, and must sign IRB-approved consent form indicating such understanding.
* Life-expectancy at least 12 months
* Patients currently receiving a second-generation androgen receptor (AR) inhibitor (e.g. enzalutamide, abiraterone, darolutamide, apalutamide) and must have had 1) PSA decline on treatment and 2) now have PSA increase over nadir while still on treatment (patients must be registered within 12 weeks of first documented PSA increase) (ACQUIRED RESISTANCE COHORT ONLY)

Exclusion Criteria:

* Must not have uncontrolled diabetes (fasting blood sugar > 200 mg/dL or inability to safely hold diabetes medication or fast 6 hours prior to FDG PET scan)
* Prior treatment with second-generation AR inhibitor for prostate cancer in the metastatic disease setting (prior second-generation AR inhibitor in the neoadjuvant or adjuvant setting is permitted unless patient developed progression while on treatment) (INTRINSIC RESISTANCE COHORT, AR-INHIBITOR GROUP ONLY)
* Pain or clinical symptoms from metastatic prostate cancer requiring opioid analgesics
* Known neuro-endocrine prostate cancer
* Prior radioisotope therapy for castration-resistant prostate cancer
* To avoid the possibility of unintended coercion, vulnerable populations such as incarcerated subjects, subjects unable to provide their own informed consent and non-English speaking patients will not be considered

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men of all races and ethnic groups are eligible for this trial. Women are excluded given that prostate cancer is a male disease.
Enrollment: 20 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Characterize intrinsic resistance based on FDG and PSMA PET through change in individual lesion update levels. | Baseline to 12 weeks
  Changes in individual lesion update levels (ΔiSUVtotal) will be calculated. SUVtotal is a metric of activity, for which less activity is better.
Characterize change in intrinsic resistance based on FDG and PSMA PET. | Baseline to 12 weeks
  Changes in individual lesion update levels (ΔiSUVtotal) will be calculated. SUVtotal is a metric of activity, for which a decrease in activity is better.
Characterize change in intrinsic resistance based on FDG and PSMA PET. | 12 weeks to 36 weeks
  Changes in individual lesion update levels (ΔiSUVtotal) will be calculated. SUVtotal is a metric of activity, for which a decrease in activity is better.
Characterize change in intrinsic resistance based on FDG and PSMA PET. | Baseline to 36 weeks
  Changes in individual lesion update levels (ΔiSUVtotal) will be calculated. SUVtotal is a metric of activity, for which a decrease in activity is better.
Characterize acquired resistance at the time of progression | Baseline to 36 weeks
  Percentage and absolute changes in individual lesion update levels (ΔiSUVtotal) will be calculated.

SECONDARY OUTCOMES:
Correlate amount of intrinsic resistance on FDG and PSMA PET to predict time to PSA progression | Baseline to 36 weeks
  Analysis will be conducted to evaluate whether changes in lesion uptake values predict time to PSA progression. PSA progression will be 25% increase and >2 ng/mL above PSA nadir
Correlate amount of intrinsic resistance on FDG and PSMA PET to predict time to radiographic progression | Baseline to 36 weeks
  Analysis will be conducted to evaluate whether changes in lesion uptake values predict time to radiographic progression. Time to radiographic progression will be defined as the number of days to confirmed radiographic progression using Prostate Cancer WorkingGroup 3 (PCWG3) criteria.
Correlate amount of intrinsic resistance on FDG and PSMA PET to predict time duration on treatment | Up to 36 weeks
  Analysis will be conducted to evaluate whether changes in lesion uptake values predict duration of treatment. Duration of treatment will be defined as the time from treatment start, to treatment discontinuation (and reason for discontinuation) using PCWG3 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Liu, MD, Principal Investigator — University of Wisconsin, Madison; Robert Jeraj, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No